CLINICAL TRIAL: NCT04480164
Title: A Randomized Double-blind Ascending-dose Placebo-controlled Study of N-desmethylclobazam in Patients With Peripheral Neuropathic Pain
Brief Title: Evaluation of the Safety and Efficacy of N-desmethylclobazam in Patients With Peripheral Neuropathic Pain
Acronym: NDMC-201
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment rate and end of study finding
Sponsor: Besson Marie (Other)
Responsible Party: Sponsor-Investigator, Besson Marie, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-01113
Record Dates: First submitted 2020-06-11; First posted 2020-07-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: 3 Sequences separated by 2 interim analyses evaluating safety and PK linearity. Sequence 1: 8 Patients randomized to placebo or NDMC 40mg/day (ratio 1:3) qd for 6 weeks. Sequence 2 will be initiated following the first interim analysis.
  Sequence 2: 8 Patients randomized to placebo or NDMC 60mg/day (ratio 1:3) qd for 6 weeks. Sequence 3 will be initiated following the second interim analysis. Otherwise Sequence 2 will be extended to a total of 30 placebo and 32 patients.
  Sequence 3: 60 Patients randomized to placebo or NDMC 60mg/day (ratio 28:32) bid for 6 weeks. Patients who do not tolerate 120mg/day will be authorized to step down to 60mg/day during the up titration period.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NDMC 40 mg/day (Experimental): Oral administration of two NDMC 20mg capsules per day over 6 weeks
  Interventions: Drug: NDMC
- NDMC 60 mg/day (Experimental): Oral administration of three NDMC 20mg capsules per day over 6 weeks
  Interventions: Drug: NDMC
- NDMC 120 mg/day (Experimental): Oral administration of six NDMC 20mg capsules per day over 6 weeks
  Interventions: Drug: NDMC
- Placebo (Placebo Comparator): Oral administration respectively, according to the experimental arm considered, of two, three or six placebo capsules per day over 6 weeks
  Interventions: Drug: NDMC

INTERVENTIONS:
Drug: NDMC — Repeated oral administration of ascending daily doses of NDMC (40mg, 60mg,120mg/day) vs placebo in 3 sequential cohorts
  Other Names: Placebo

SUMMARY:
Neuropathic pain (NP) affects up to 8% of the general population and its successful management is an unmet medical need. Half of the patients report inadequate response to therapy and unwanted side effects such as sedation and cognitive impairments, limiting drug use in daily practice and significantly accounting for the high incidence of treatment failure. Dysfunction of synaptic inhibition within the spinal cord is known to be one of the main contributing factors to central sensitization that governs NP. Facilitation of GABAergic inhibition in the dorsal horn through GABAA receptors allosteric modulation would be a rational approach to NP management. New insights on the associations between GABAA receptors α subunits and function have opened new perspectives in preclinical research. Data from genetically modified mice demonstrates the possibility, through selective allosteric modulation of the GABAA receptor, to induce its beneficial antihyperalgesic effects without inducing its cognitive and sedative effects. N-Desmethylclobazam (NDMC), clobazam's main active metabolite, demonstrated in vitro and in vivo a high selectivity profile with a clear preference for GABAA α2-subtypes receptors (antihyperalgesia) over α1 receptors responsible for sedative effects across a wide concentration range. Taking into consideration the high prevalence and burden of neuropathic and chronic pain worldwide and the fact that these patients are nowadays left with sedative and only partially effective drugs, NDMC qualifies as a good molecule to seek confirmation of the clinical utility of selective GABAA allosteric modulators in NP patients.The main objective is to assess the efficacy of repeated doses of NDMC on neuropathic pain compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix 1: Informed Consent Form);
* Male or female participants (if female: post-menopausal or surgically sterile, or using a highly effective method of contraception);
* Between 18 and 85 years of age;
* Body mass index ≥ 18 and < 40 (kg/m2);
* Patients diagnosed with small fiber neuropathy OR suffering from peripheral neuropathic pain related to diabetic peripheral neuropathy; post-herpetic neuralgia; HIV-associated neuropathic pain; post-traumatic/postoperative peripheral neuropathy; chemotherapy associated peripheral neuropathy or nerve root/medullar compression with sensory/motor deficit OR presenting with neuropathic pain associated with diagnosed rare hereditary or acquired neurological disease; AND who presented insufficient response to at least one attempt with one of the currently recommended pharmacological treatment for neuropathic pain taken at efficacious dose OR who have interrupted treatment because of tolerance issue OR who have previously declined pharmacological pain management;;
* Pain duration for at least 3 months;
* Preceding week pain recall score ≥ 4 on NRS Scale;
* Score ≥ 4 on DN4 questionnaire;
* Willing to withdraw from prohibited medications;
* Poor-metabolizers (PM) for CYP2C19 are only eligible for Sequence 3

Exclusion Criteria:

* Contraindications to benzodiazepines.(including known hypersensitivity reaction)
* Women who are pregnant or breast feeding or who intend on becoming pregnant during the course of the study;
* Woman of childbearing potential, not using and not willing to continue using a highly effective method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases;
* Abnormal ASAT or ALAT plasma levels (> 3x ULN);
* Reduced renal function (GFR < 60 mL/min/1.73m2);
* Changes in existing (or addition of new) concomitant interventional pain management (including local anaesthetic infiltration, local nerve block, central neurostimulation therapy) and other non-pharmacological intervention such as desensitization techniques, acupuncture, transcutaneous electrostimulation, hypnosis;
* Co-existing nociceptive or inflammatory aetiology to the current pain symptoms;
* Unable to withdraw from prohibited medications before randomization;
* Epilepsy;
* History of drug, alcohol or substance abuse in the past 5 years (with the exception of stable opioid substitution therapy in the past 5 years);
* Current unstable psychiatric disorder or any such disorder that may impair patient's abilities to follow study procedures;
* Sleep apnea (unless treated with CPAP with an oxygen desaturation index < 5 per hour), myasthenia gravis, severe respiratory failure;
* Participation in another study with investigational drug within the 3 month preceding and during the present study (a wash-out of period at least 3 months is necessary prior to screening).
* Score < 24 on MMS in patients over 65 years of age

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Weekly Average of daily Pain intensity score (WAP) | Week 0, Week 6 following first drug administration
  Participant will self-rate once every day his average daily pain. The weekly average of daily pain intensity score will be derived from the 7 (at least 5) recordings preceding Baseline (Week 0) and Final evaluation (Week 6). Numerical Rating Scale = 0 "no pain" to 10 = "worst possible pain". The primary outcome will be the change from Baseline to Final evaluation.

SECONDARY OUTCOMES:
Evolution of Weekly Average of daily Pain intensity score (EWAP) | Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 following first drug administration
  Assessment of the evolution overtime of the weekly average of daily pain intensity score between Baseline (Week 0) and Final evaluation (Week 6).
Weekly Average of daily subjective feeling of Sedation (WAS) | Week 0, Week 6 following first drug administration
  Participant will self-rate once every day his daily subjective feeling of sedation. The weekly average of daily subjective feeling of sedation score will be derived from the 7 (at least 5) recordings preceding Baseline (Week 0) and Final Evaluation (Week 6). Numerical Rating Scale = 0 "not sleepy" to 10 = "extremely sleepy".
Evolution of Weekly Average of daily subjective feeling of Sedation (EWAS) | Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 following first drug administration
  Assessments of the evolution overtime of the weekly average of daily subjective feeling of sedation score, each week between Baseline (Week 0) and Final evaluation (Week 6).
Composite 2-Dimension Score (C2-D) | Week 0, Week 6 following first drug administration
  The Composite 2-Dimension score will assess the benefit/tolerance balance of NDMC for each dose. The score is defined as the aggregated value of the changes between baseline and final evaluation on the weekly average of daily pain intensity score and the weekly average of daily subjective sedation score. Score ranges from -10 to + 16. Score ≤ -2 indicates a favorable balance and score ≥ 2 an unfavorable balance.
Evolution of Composite 2-Dimension Score (EC2-D) | Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 following first drug administration
  Assessments of the evolution overtime of the Composite 2-Dimension score, each week between Baseline (Week 0) and Final evaluation (Week 6).
Douleur neuropathique 4 questionnaire (DN4) | Week 0, Week 2, Week 6 following first drug administration
  Participant will complete the DN4 questionnaire which is a screening tool for neuropathic pain consisting of interview questions. This questionnaire gives a score ranging from 0 (better) to 10 (worse); a score ≥4 is an indicator of plausible neuropathic pain.
Neuropathic Pain Symptom Inventory (NPSI) | Week 0, Week 2, Week 6 following first drug administration
  Participant will complete the NPSI questionnaire which is an inventory tool for neuropathic pain consisting of interview questions.This questionnaire has 12 scaled scores and gives a score ranging from 0 (better) to 100 (worse)
Short Form Questionnaire (SF-36) | Week 0, Week 2, Week 6 following first drug administration
  Participant will complete the health status questionnaire consisting of 36 interview questions. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
Hospital Anxiety and Depression Scale (HADS) | Week 0, Week 2, Week 6 following first drug administration
  Participant will complete the anxiety and depression questionnaire consisting in two sets of 7 questions on anxiety or depression. HADS gives anxiety and depression scores both ranging from 0 (better) to 21 (worse)
Patient Global Impression of Change (PGIC) | Visit 1 to Visit 7
  Participant will complete the PGIC questionnaire, which is a 7-point scale ranging from -3 (very much worse), 0 (no change), to +3 (very much improved) answering the question: "Please, indicate how you feel now, compared to how you felt before receiving treatment in this study"
Clinician Global Impression of Improvement (CGI-I) | Week 0, Week 2, Week 6 following first drug administration
  Investigator will complete CGI questionnaire which is a 7-point CGI scale: from 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse) to 7 (very much worse) answering the question: "Please, indicate how much the patient's condition has improved or worsened relative to a baseline state at the beginning of the intervention"
Medical Outcome Study Sleep Score (MOS-Sleep) | Week 0, Week 2, Week 6 following first drug administration
  Participant will complete the MOS-sleep questionnaire, which is composed of 12 items. Higher scores reflect more of the attribute implied by the scale names
Responder Rates (30% / 50%) | Week 0, Week 6 following first drug administration
  Participants will be dichotomized into "responders" and "non-responders" categories. These transformations will be based on the reduction of at least 30%, respectively 50%, of the weekly average daily pain intensity score between Baseline (Week 0) and Final evaluation (Week 6).
Rescue Medication Rate | Week 0, Week 6 following first drug administration
  Participants will be dichotomized into "rescue med" and "no rescue med" categories. This transformation will be based on the use of rescue medications between Baseline (Week 0) and Final evaluation (Week 6).
Withdrawal Rate | throughout the study (up to 6 weeks)
  Participants will be dichotomized into "early withdrawal" and "completion" categories. This transformation will be based on the occurrence of premature withdrawal related to lack of efficacy or due treatment emergent adverse effect between Baseline (Week 0) and Final evaluation (Week 6).

OTHER OUTCOMES:
Steady state NDMC Cmin concentration | Week 0, Week 2, Week 6 following first drug administration
  Determination of mean NDMC Cmin concentrations at steady state following daily administration (40mg, 60mg, 120mg) in 3 sequential cohorts of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Besson, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No